CLINICAL TRIAL: NCT03262194
Title: Relevance of Gastric Aspirate in HCMV Detection
Acronym: VIRULAG
Status: Terminated | Type: Observational
Why Stopped: The introduction of new recommendations for early neonatal infection has drastically reduced the need for gastric aspiration at birth.
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2017/314
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Cytomegalovirus Infections; Hypotrophic Newborns
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Human cytomegalovirus (CMV) is the leading cause of neonatal viral infection and can have a significant impact on the neurosensory development of newborns and especially premature infants. CMV infection can result from materno-fetal transmission during pregnancy (congenital infection) or postnatal transmission. The prevalence of congenital CMV infection in the newborn is estimated to be between 0.1 and 0.5%. Among the newborns in utero infected by CMV, it is estimated that 10-15% will present symptoms at birth (hypoacousia / unilateral or bilateral deafness, microcephaly, chorioretinitis, psychomotor retardation, etc.) and 0.5% of them will die. 20% of infected infants, mainly symptomatic newborns, suffer permanent sequelae, mainly loss of hearing. Many asymptomatic children at birth will present hearing loss and other delayed neurological complications. A progressive neurosensory hearing loss may develop for 13-15% of asymptomatic newborns at birth. Deafness is bilateral in 50% of cases, severe in more than 50% of cases, and its occurrence is often delayed. The hearing loss has a significant impact on the future life of the child, mainly on language acquisition and school performance.

A systematic CMV screening is not currently recommended at birth due to the frequency of asymptomatic forms, difficulty in fetal diagnosis and prognosis, lack of consensus for preventive and curative treatment of the infection. New treatments are being evaluated and encouraging results could revive the debate.

PCR from urine is the gold standard for the diagnosis of CMV infection. Urine collection is not systematic in newborns and its realization can sometimes be difficult. On the other hand, in children at risk (hypotrophy, prematurity, infectious risks, fetal distress or respiratory distress at birth), gastric aspiration is systematically performed at birth to overcome obstruction of the upper aero-digestive tract, to prevent oesophageal atresia, to avoid inhalation by reflux and sometimes to make a bacteriological diagnosis.

Our hypothesis is that this liquid could be used for the detection of CMV infection without adding any invasive action in newborns. Ultimately, gastric aspirate could allow for routine CMV screening in children at risk and thus allow for appropriate care by nursing staff.The occurrence of immediate or delayed sensory sequelae in these children would be then limited.

ELIGIBILITY:
Inclusion Criteria of the newborn:

- Child born in maternity and / or child hospitalized in the Neonatal Médicine Department of the University Hospital of Besançon for which a urine sample (minimum volume = 0.5 mL) and a gastric aspiration fluid sample (minimum volume = 0.7mL) were collected (regardless of gender, birth weight or pathology presented at admission).

Exclusion Criteria of the newborn:

* Child died before the sampling
* A volume of gastric aspiration fluid dedicated to the study less than 0.7 mL.
* An impossible collection of urine (malformation, skin irritation of the perineum, contamination with meconium).

Ages: 1 Minute to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hypotrophic newborns
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Match between gastral aspirate PCR results and urine PCR results | day 7
  Match between gastral aspirate polymerase chain reaction results and urine polymerase chain reaction results

CONTACTS AND LOCATIONS:
Overall Officials: Thiriez Gérard, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- Chu Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No